CLINICAL TRIAL: NCT04285268
Title: A Phase 2 Study of Rituximab, Venetoclax (ABT 199) and Bortezomib in Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Rituximab, Venetoclax, and Bortezomib for the Treatment of Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was never submitted to the IRB for review and approval.
  No research subjects were enrolled.
  .
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, CINJRegulatory, CINJ Regulatory - The PI is no longer affiliated with Rutgers, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011915; NCI-2020-00904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 011915 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent Burkitt Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory Burkitt Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib; Rituximab; CT-P10; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (rituximab, venetoclax, bortezomib) (Experimental): Patients receive rituximab IV on day -1 of cycle 1, then on day 1 of cycles 2-6. Patients also receive venetoclax PO QD on days 1-14 and bortezomib IV or SC on day -1 of cycle 1, then on days 1, 8, and 15 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles for rituximab and up to 26 cycles for venetoclax and bortezomib in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Rituximab; Drug: Venetoclax

INTERVENTIONS:
Drug: Bortezomib — Given IV or SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well rituximab, venetoclax, and bortezomib work in treating patients with diffuse large B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Venetoclax and bortezomib may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. Giving rituximab, venetoclax, and bortezomib may slow or stop the growth of cancer cells in patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) of rituximab, venetoclax, and bortezomib in relapsed/refractory diffuse large B-cell lymphoma.

SECONDARY OBJECTIVES:

I. To describe the safety profile of rituximab, venetoclax, and bortezomib in diffuse large B-cell lymphoma (DLBCL).

II. To describe the progression free survival of subjects enrolled to the study.

III. To describe the median overall survival of subjects enrolled to the study. IV. To describe the complete remission (CR) rate, the partial remission (PR) rate and the duration of response (DoR) of rituximab, venetoclax, and bortezomib in relapsed/refractory DLBCL.

EXPLORATORY OBJECTIVE:

I. To describe the association of BCL2 expression status, measured by immunohistochemistry (IHC), with ORR, CR and PR rates.

OUTLINE:

Patients receive rituximab intravenously (IV) on day -1 of cycle 1, then on day 1 of cycles 2-6. Patients also receive venetoclax orally (PO) once daily (QD) on days 1-14 and bortezomib IV or subcutaneously (SC) on day -1 of cycle 1, then on days 1, 8, and 15 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles for rituximab and up to 26 cycles for venetoclax and bortezomib in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory DLBCL defined as any of the following:

  * Confirmed DLBCL/Burkitt lymphoma (BL)/B-cell lymphoma, unclassifiable (BCLU) by World Health Organization (WHO) 2016 classification
  * Double hit lymphoma (DHL) phenotype as confirmed by FISH (fluorescent in-situ hybridization) or IHC (immunohistochemistry)
* Relapsed or progression of disease after at least one prior line of standard rituximab-cyclophosphamide-hydroxydaunorubicin-oncovin-prednisone (R-CHOP), rituximab-etoposide-prednisone-oncovin-cyclophosphamide-hydroxydaunorubicin (R-EPOCH) or other R-CHOP-like therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* No prior treatment with a proteasome inhibitor or prior BCL2 inhibitor
* No cytotoxic chemotherapy within 2 weeks prior to study treatment
* Patients who are not candidates for salvage stem cell transplant or patients who are not candidates for CAR-T (chimeric antigen receptor T-cell) therapy, patients who have progressed or relapsed after a salvage transplant or CAR-T therapy are eligible
* Patients must give informed consent
* Prior radiation therapy allowed to < 25% of the bone marrow and patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Patients treated with standard postoperative adjuvant radiation therapy for other cancers are allowed. Prior radiotherapy must be completed 14 days before study entry. Lesions that have been radiated in the advanced setting cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy
* Patients with lower blood counts due to marrow involvement by DHL will be eligible for the study
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 50,000/uL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 X institutional upper limit of normal (ULN)
* Creatinine < 1.5 the upper limit of normal

Exclusion Criteria:

* Patients who have had prior proteasome inhibitor therapy or prior therapy with venetoclax
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Serious concomitant systemic disorders (including active infections) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Patients with history of hepatitis B with negative viral load are eligible (including latent carriers and patient with history of active disease who required treatment)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to venetoclax and bortezomib or other agents used in the study
* Subjects with human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS) which is not well controlled on antiviral therapy
* Patients who have received autologous hematopoietic stem cell transplantation within 12 months
* Subject has received the following within 7 days prior to the first dose of study drug: Steroid therapy for anti-neoplastic intent, strong and moderate CYP3A inhibitors and/or strong and moderate CYP3A inducers
* The effects of combination venetoclax and bortezomib may cause fetal harm. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 12 weeks after. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-06 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  Defined as the proportion of subjects who achieve a best response of a partial response (PR) or better. The ORR (complete and partial responses) will be reported as a percentage with a 95% confidence interval. If response is missing for any patients, those patients will still be included in the denominator when reporting the response rate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post treatment
  Toxicity parameters will be defined by National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (V) 5.0. Descriptive statistics will be provided for the safety data.
Progression free survival (PFS) | From study enrollment to disease progression or death from any cause, assessed up to 4 years
  The Kaplan-Meier curve will be used to estimate the corresponding PFS distribution and median PFS for patients treated on this study.
Overall survival (OS) | From study enrollment to the date of death from any cause, assessed up to 4 years
  The Kaplan-Meier curve will also be used to estimate the corresponding OS distribution and median OS for all treated patients. If a subject has not died, their survival time will be censored at the date of last contact ("last known alive date").
Complete response (CR) and partial response (PR) rates | Up to 4 years
  Defined as the proportion of subjects who achieve a best response of CR or PR respectively.
Duration of response (DoR) | From when measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 4 years
  The Kaplan-Meier curve will be used to estimate the corresponding DoR distribution and median DoR for patients treated on this study who achieve a CR or PR.

OTHER OUTCOMES:
BCL2 protein expression | Up to 4 years
  BCL2 protein expression by immunohistochemistry will be defined as positive or negative based on the most recent available biopsy report of each patient's diffuse large B-cell lymphoma. Descriptive statistics will be provided for the exploratory analysis of BCL2 expression and response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Bannerji, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States